CLINICAL TRIAL: NCT01297218
Title: Open-Label, Single-Center, Phase 1 Clinical Trial to Evaluate the Safety and the Efficacy of NEUROTSTEM®-AD in Patients With Dementia of the Alzheimer's Type
Brief Title: The Safety and The Efficacy Evaluation of NEUROSTEM®-AD in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-CR-007
Record Dates: First submitted 2011-02-11; First posted 2011-02-16 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Dementia of the Alzheimer's Type
Keywords: Alzheimer, Mesenchymal Stem Cells, Umbilical Cord Blood
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NEUROSTEM®-AD (Experimental)
  Interventions: Biological: Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells — DOSE A - 250,000 cells per 5 uL per 1 entry site, 3 million cells per brain DOSE B - 500,000 cells per 5 uL per 1 entry site, 6 million cells per brain
  Other Names: NEUROSTEM®-AD

SUMMARY:
The primary purpose of this study is to evaluate the safety and the tolerability of NEUROSTEM®-AD (Human Umbilical Cord Blood Derived Mesenchymal Stem Cells) and to assess the maximum tolerated dose (MTD). This study is also to investigate the efficacy of this study drug in patients with dementia of Alzheimer's type.

DETAILED DESCRIPTION:
Most of the treatments for Alzheimer disease are chemical drug that is designed to temporarily increase acetylcholine, based on the cholinergic hypothesis. These drugs can improve the symptoms but is not able to inhibit the disease progression. New drugs from the disease have been developed but they have not been successful yet.

Mesenchymal stem cells (MSC) are capable of differentiating into various tissues. Due to the characteristics of the cells it has been widely investigated in tissue regeneration. In addition, the paracrine effect of MSC in microenvironment has been recently reported. MSC has been developed as an immunomodulation cell therapy product because it has been known that it does not cause immunological rejection in allo- and xeno-transplantation. Clinical studies showed that umbilical cord blood-derived MSC is immunologically stable and not toxic.

This study is to evaluate the safety and the tolerability of NEUROSTEM®-AD (Human Umbilical Cord Blood Derived Mesenchymal Stem Cells) and to assess the maximum tolerated dose (MTD). This study is also to investigate the efficacy of this study drug in patients with dementia of Alzheimer's type.

ELIGIBILITY:
Inclusion Criteria:

* Korean men and women who are age 50 or older
* Dementia as determined by DSM-IV criteria
* Probable alzheimer's disease as determined by NINCDS-ADRDA criteria
* K-MMSE score in the range of 10 to 24
* Positive result of PIB-PET imaging (SUV > 1.5,when comparing the result for the cerebellum with the result for the frontal lobe)
* Voluntarily participating subject who sign the consent form

Exclusion Criteria:

* Subject with psychological diseases (i.e. depression, schizophrenia, bipolar disorder, etc)
* Subject with dementia caused by other than Alzheimer's disease (i.e. infection of central nervous system, Creutzfeld-Jacob disease, severe head trauma, Pick's disease, Huntington's disease, and Parkinson's disease)
* Subject with vascular dementia as determined by the clinical criteria of DSM IV and the imaging criteria of Erkinjuntii
* Subject with severe white matter hyperintensities (WMH); Severe WMH is defined that length of the deep white matter is 25 mm or longer and length of the periventricular capping/banding is 10 mm or longer.
* Subject who have had stroke in 3 months.
* Subject with liver disease (two times higher than normal range of ALT/AST)
* Subject with severe kidney failure (1.5mg/dL of serum creatinine or more)
* Pregnant women or lactating women
* Hemoglobin < 9.5g/dL for men, < 9.0 g/dL for women; Total WBC count < 3000/mm3; Total bilirubin ≥ 3 mg/dL
* Subject who is suspect to have active lung diseases, based on check X-ray result from Visit 1
* Women of childbearing age who reject to practice contraception
* Subject who have been excluded in the subject selection process for this study before
* A platelet count < 150,000/mm3; PT ≥ 1.5; INR or aPTT ≥ 1.5 X control
* Subject with cancer
* History of alcohol or drug abuse
* Subject who cannot undergo MRI, CT, or PET screening
* Subject who cannot undergo anesthesia or stereotactic brain injection
* Subject who is determined inappropriate by the investigators

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse event | 12 weeks from post-administration
  Number of participants with adverse event, number of participants with normal range of vital signs, mixed lymphocyte reaction, and laboratory examination

SECONDARY OUTCOMES:
Changes from the baseline in ADAS-cog at 12 weeks post-dose | 12 weeks from post-administration
  Changes from the baseline in ADAS-cog, S-IADL, K-MMSE, CGA-NPI, ADAS-Cog, serum transthyretin, amyloid beta and tau in cerebrospinal fluid, PIB-PET and FDG-PET at 12 weeks post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Duk L. Na, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Seo SW, Chang JW, Lee JI, Kim CH, Chin J, Choi SJ, Kwon H, Yun HJ, Lee JM, Kim ST, Choe YS, Lee KH, Na DL. Stereotactic brain injection of human umbilical cord blood mesenchymal stem cells in patients with Alzheimer's disease dementia: A phase 1 clinical trial. Alzheimers Dement (N Y). 2015 Jul 26;1(2):95-102. doi: 10.1016/j.trci.2015.06.007. eCollection 2015 Sep. PMID 29854930